CLINICAL TRIAL: NCT05641142
Title: Prospective Study of Antiplatelet and Anticoagulation Therapy in Hereditary Haemorrhagic Telangiectasia
Acronym: PROPLACO-Tel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RBHP 2022 GROBOST; 2022-A00754-39 (Other: 2022-A00754-39)
Record Dates: First submitted 2022-11-18; First posted 2022-12-07 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Rendu Osler Disease
Keywords: epistaxis; hemorrhage; anticoagulant therapy; antiplatelet therapy
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis; Hemorrhage

STUDY DESIGN:
Intervention Model Description: cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort study (Other): a single arm, the anticoagulant and/or antiplatelet treatment is not conditioned by the study
  Interventions: Other: monitoring the use of anticoagulant and/or antiplatelet therapy in patients with osler rendering disease

INTERVENTIONS:
Other: monitoring the use of anticoagulant and/or antiplatelet therapy in patients with osler rendering disease — Monitoring:
  * hemoglobin and ferritin levels
  * transfusion or intravenous iron
  * hospitalization for bleeding or thrombose
  * digestive bleeding and/or another haemorrhagic accident
  * severity of epistaxis
  * quality of life

SUMMARY:
The goal of this clinical trial is to evaluate in real life, in patients with Hereditary Hemorrhagic Telangiectasia (HHT), the tolerance of the strategy of use of anticoagulant and/or antiplatelet, by comparing a new exposure period (first trimester of treatment) to a period of reference non-exposure (last trimester before start of treatment).

DETAILED DESCRIPTION:
Currently there are no recommendations on the use of anticoagulant and/or antiplatelet treatment in patients with Rendu-Osler Disease.

The main question this study aims to answer is:

• to better determine which anticoagulant and/or antiplatelet therapy are best tolerated or if they are equivalent in Rendu-Osler disease because this type of treatment is often used in urgent and/or vital situations.

Participants will have a 2-year follow-up with biological monitoring of ferritin and hemoglobin level and ESS (Epistaxis Severity Score) and QoL-HHT (Quality of Life Hereditary Hemorrhagic Telangiectasia) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Rendu-Osler disease with an indication of antiplatelet and/or anticoagulant introduced for less than 3 months (inclusion period within 3 months of exposure)
* Age > 18 years old
* Patient able to understand and agree to participate in the study
* Affiliation to a social security system

Exclusion Criteria:

* Patient with an indication of antiplatelet and/or anticoagulant but for whom treatment has not been introduced or introduced for more than 3 months
* Refusal to participate
* Pregnant woman or who are breast feeding
* Patients under maintenance of justice, wardship or legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Number of transfusions and/or intravenous iron | 3 months after exposure to anticoagulants and/or antiplatelet
  Number of transfusions and/or intravenous iron before (3 months) and within 3 months after exposure to anticoagulants and/or antiplatelet in patients with Rendu-Osler disease.

SECONDARY OUTCOMES:
Biological parameters | 3 months after exposure to anticoagulants and/or antiplatelet
  Evolution of ferritin levels.
Biological parameters | 3 months after exposure to anticoagulants and/or antiplatelet
  Evolution of hemoglobin levels.
Bleeding | 3 months after exposure to anticoagulants and/or antiplatelet
  Onset of digestive bleeding and/or occurrence of a new hemorrhagic accident or major hemorrhagic event and/or hospitalisation for hemorrhage.
Anticoagulant and/or antiplatelet treatment | week 104 after patient inclusion
  Frequency of continuation and/or modification and/or cessation of treatment if indication maintained.
Thrombotic accident | week 104 after patient inclusion
  Frequency of occurrence of a new arterial and/or venous thrombotic accident and/or death
Epistaxis | week 12, 52 and 104 after patient inclusion
  Evolution of epistaxis severity via ESS score
Evaluation of Quality of life | week 6, 12, 52 and 104 after patient inclusion
  Quality of life assessment via QoL-HHT questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GROBOST, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (18):
- France (18):
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU de Caen Normandie, Caen
  - CHU clermont-ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHRU de Lille, Lille
  - Hospices Civiles de Lyon, Lyon
  - Assistance Publique - Hôpitaux de Marseille, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - AP-HP - Hôpital Ténon, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHRU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse